CLINICAL TRIAL: NCT02641951
Title: Stellate Ganglionic Block Versus Combined Stellate Ganglionic Block and Modified Pectoral Nerve Block in Treatment of Post Mastectomy Pain Syndrome.
Brief Title: Stellate Ganglionic Block Versus Stellate Ganglionic Block Plus Pecs II Block for Mastectomy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R/15.08.41
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Post Mastectomy Pain Syndrome; After Breast Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stellate ganglionic block (Placebo Comparator): Ultrasound guided stellate ganglionic block
  Interventions: Other: Stellate ganglionic block
- Pecs II block (Active Comparator): Ultrasound guided Pecs II block
  Interventions: Other: Pecs II block

INTERVENTIONS:
Other: Stellate ganglionic block — Ultrasound guided stellate ganglionic block
  Arms: Stellate ganglionic block
Other: Pecs II block — Ultrasound guided Pecs II block
  Arms: Pecs II block

SUMMARY:
Post mastectomy pain syndrome result from surgical damage to the intercostobrachial nerve, the lateral cutaneous branch of the second intercostal nerve that is often resected at mastectomy. result from surgical damage to the intercostobrachial nerve, the lateral cutaneous branch of the second intercostal nerve that is often resected at mastectomy, A second version of the pectoral nerve block is described, called ''modified Pecs block'' or Pecs block type II.

This novel approach aims to block at least the pectoral nerves, the intercostobrachial, intercostals III-IV-V-VI and the long thoracic nerve. These nerves need to be blocked to provide complete analgesia during breast surgery

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of ultrasound guided stellate ganglionic block alone versus stellate ganglionic block plus pecs II block in management of chronic postmastectomy pain ,patient will be trained to use visaual analog scale to describe their pain range of movement will be assessed using manual geniometry at post procedure visits at one month ,3 months and 6 months procedures in each group will done using ultrasound guidance mixture will be used.

All patients will be informed about the procedure and its possible consequences after detailed explanation of protocol of this study. Written informed consents will be obtained before the procedure.

With each block, an intravenous cannula will be inserted and secured. All suitable resuscitation equipment and drugs will be available. Vital signs (heart rate, blood pressure, and oxygen saturation) will be monitored throughout the procedure and up to 1 hour after the block performance. Midazolam 0.02 ug/kg will be administered intravenously as premedication.

Brief evaluation will be done for all patients with regard to their systemic diseases, general condition, and coagulation status.

All patients will be familiar with the use of 10-cm visual analogue scale score (VAS) identifying 0 as no pain and 10 as worst imaginable pain.Basal assessment of range of movement for abduction ,external rotation ,and forward flextion using manual geniometry and patients will be asked to complete Quality of life questionnaire

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status III or IV.
* Patients having irradiating pain of anterior chest wall and axilla after breast surgery.
* Patients having irradiating pain of ipsilateral arm after breast surgery
* Pain not responding to conservative treatment
* Pain persisting for more than 3 month

Exclusion Criteria:

* Local skin infection
* Coagulation or blood disease
* Pregnancy
* Postpartum or lactating females
* Allergy to the study medications.
* Severely altered consciousness level.
* Psychiatric disorder
* Drug abuse
* Spine or chest wall deformities

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Pain scores | for six months after the procedure
  100 mm- visual analog pain scale

SECONDARY OUTCOMES:
The range of motion of the glenohumeral joint | for six months after the procedure
  Improvements in the range of motion of the glenohumeral joint, which included forward extension and external rotation will be recorded using scoring system score 0 to 9 for some movements range and 0 to 160 for others
The quality of life score | for six months after the procedure
  The quality of life will be assessed using the score QOLSF 36

CONTACTS AND LOCATIONS:
Overall Officials: Zenat E Mohamed, MD, Study Chair — Department of Anaesthesia, Surgical Intensive Care and Pain Medicine, College of Medicine, Mansoura University, Mansoura, Egypt; Reem A Sharkawy, MD, Study Director — Department of Anaesthesia, Surgical Intensive Care and Pain Medicine, College of Medicine, Mansoura University, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: Undecided